CLINICAL TRIAL: NCT01802398
Title: Improving Syncope Risk Stratification in Older Adults
Acronym: SRS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Benjamin Sun, M.D., Associate Professor, Emergency Medicine, University of Pennsylvania
Other Study IDs: NIH R01 HL111033-01A1
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Syncope
Keywords: Risk Stratification; Syncope; Geriatric
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be collected for standardized cardiac biomarker testing. Samples will be split into two aliquots for testing and long-term storage. Aliquots in long-term -80˚C storage will be used for future studies of novel tests.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Observational cohort study of older (age≥60 years) adults who present to an emergency department with syncope (otherwise known as fainting)

SUMMARY:
Syncope (temporary loss of consciousness) is a frequent reason for an emergency department (ED) visit among older adults. The current ED evaluation of syncope frequently leads to hospitalization, results in low diagnostic yield, and is enormously costly. The purpose of this protocol is to improve risk prediction for syncope. Improved risk prediction will inform the design of interventions to safely reduce unnecessary health service use.

This is a multi-center, prospective, observational cohort study of older (age≥60 years) adults who present to an emergency department with syncope (otherwise known as fainting). The primary outcome is a composite of 30-day cardiac death and serious cardiac events.

Study Aims and Hypotheses are:

Specific Aim 1. Describe serious outcomes after unexplained syncope; rates and reasons for admission; and frequency, diagnostic yield, and therapeutic impact of inpatient diagnostic tests.

H1: Current patterns of care representing a diversity of practice settings and patient populations are costly with low clinical benefit.

Specific Aim 2. Derive and validate a novel risk prediction model for 30-day cardiac death and serious cardiac outcomes after unexplained syncope.

H2: Explicit criteria including contemporary cardiac biomarkers will improve risk stratification compared to unstructured physician assessment and published risk models.

Specific Aim 3. Assess safety and costs of a risk-tailored diagnostic algorithm compared to existing care for unexplained syncope.

H3: A risk-tailored diagnostic algorithm can safely reduce the costs of evaluating unexplained syncope in older adults.

ELIGIBILITY:
Inclusion Criteria:

1. age≥60 years; AND
2. a complaint of syncope or near-syncope. Syncope is defined as a transient loss of consciousness (LOC), associated with loss of postural tone, with immediate, spontaneous, and complete recovery. Near-syncope is the sensation of imminent syncope without loss of consciousness.

Exclusion Criteria:

* Seizure as presumptive cause of LOC
* Stroke or transient ischemic attack as presumptive cause of LOC
* LOC AFTER head trauma Confusion from baseline mental status
* Intoxicated (alcohol or other drugs)
* Medical or electrical intervention to restore consciousness
* Hypoglycemia as presumptive cause of LOC
* inability to provide follow-up information, including patients who do not speak English (or Spanish, if applicable for study site), lack phone access, or lack a permanent address
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Departments (ED)
Sampling Method: Non-Probability Sample
Enrollment: 3707 (Actual)
Dates: Start 2013-04; Primary Completion 2016-09-21 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Combined death and serious cardiac events | 30 days
  This aim tests the hypothesis that current patterns of care are costly with low clinical benefit. We will generate tables that describe the demographics, clinical characteristics, and disposition of the study cohort, stratified by occurrence of the primary outcome. Outcomes experienced by the study cohort will be described in detail.

OTHER OUTCOMES:
Non-cardiac serious events | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin C Sun, MD, Principal Investigator — Oregon Health and Science University
Locations (10):
- United States (10):
  - University of California, Davis | UC Davis, Sacramento, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Health System, Royal Oak, Michigan
  - URMC, Emergency Department, Rochester, New York
  - Wakeforest, Department of Emergency Medicine, Winston-Salem, North Carolina
  - Summa Health System, Department of Emergency Medicine (Research), Akron, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Zimmermann T, du Fay de Lavallaz J, Walter JE, Strebel I, Nestelberger T, Joray L, Badertscher P, Flores D, Widmer V, Geigy N, Miro O, Salgado E, Christ M, Cullen L, Than M, Martin-Sanchez FJ, Di Somma S, Peacock WF, Keller D, Costabel JP, Wussler DN, Kawecki D, Lohrmann J, Gualandro DM, Kuehne M, Reichlin T, Sun B, Mueller C; BASEL IX and SRS Investigators. Development of an electrocardiogram-based risk calculator for a cardiac cause of syncope. Heart. 2021 Nov;107(22):1796-1804. doi: 10.1136/heartjnl-2020-318430. Epub 2021 Jan 27. PMID 33504514
- [Derived] Probst MA, Gibson T, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Hollander JE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Risk Stratification of Older Adults Who Present to the Emergency Department With Syncope: The FAINT Score. Ann Emerg Med. 2020 Feb;75(2):147-158. doi: 10.1016/j.annemergmed.2019.08.429. Epub 2019 Oct 23. PMID 31668571
- [Derived] Probst MA, Su E, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Hollander JE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Clinical Benefit of Hospitalization for Older Adults With Unexplained Syncope: A Propensity-Matched Analysis. Ann Emerg Med. 2019 Aug;74(2):260-269. doi: 10.1016/j.annemergmed.2019.03.031. Epub 2019 May 9. PMID 31080027
- [Derived] Clark CL, Gibson TA, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Diercks DB, Hollander JE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Do High-sensitivity Troponin and Natriuretic Peptide Predict Death or Serious Cardiac Outcomes After Syncope? Acad Emerg Med. 2019 May;26(5):528-538. doi: 10.1111/acem.13709. Epub 2019 Mar 4. PMID 30721554
- [Derived] Thiruganasambandamoorthy V, Sivilotti MLA, Rowe BH, McRae AD, Mukarram M, Malveau S, Yagapen AN, Sun BC; North American Syncope Consortium. Prevalence of Pulmonary Embolism Among Emergency Department Patients With Syncope: A Multicenter Prospective Cohort Study. Ann Emerg Med. 2019 May;73(5):500-510. doi: 10.1016/j.annemergmed.2018.12.005. Epub 2019 Jan 26. PMID 30691921
- [Derived] Bastani A, Su E, Adler DH, Baugh C, Caterino JM, Clark CL, Diercks DB, Hollander JE, Malveau SE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Yagapen AN, Weiss RE, Sun BC. Comparison of 30-Day Serious Adverse Clinical Events for Elderly Patients Presenting to the Emergency Department With Near-Syncope Versus Syncope. Ann Emerg Med. 2019 Mar;73(3):274-280. doi: 10.1016/j.annemergmed.2018.10.032. Epub 2018 Dec 7. PMID 30529112
- [Derived] Chang AM, Hollander JE, Su E, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Recurrent syncope is not an independent risk predictor for future syncopal events or adverse outcomes. Am J Emerg Med. 2019 May;37(5):869-872. doi: 10.1016/j.ajem.2018.08.004. Epub 2018 Aug 24. PMID 30361153
- [Derived] Probst MA, Gibson TA, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Hollander JE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Predictors of Clinically Significant Echocardiography Findings in Older Adults with Syncope: A Secondary Analysis. J Hosp Med. 2018 Dec 1;13(12):823-828. doi: 10.12788/jhm.3082. Epub 2018 Sep 26. PMID 30255862
- [Derived] Nishijima DK, Lin AL, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Hollander JE, Nicks BA, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. ECG Predictors of Cardiac Arrhythmias in Older Adults With Syncope. Ann Emerg Med. 2018 Apr;71(4):452-461.e3. doi: 10.1016/j.annemergmed.2017.11.014. Epub 2017 Dec 21. PMID 29275946